CLINICAL TRIAL: NCT05826249
Title: A Single Center, Non-randomized, Open-label Phase I Study to Investigate the Pharmacokinetics and Safety of SIM0417/Ritonavir After Single Dose Administration in Healthy Elderly Subjects
Brief Title: Safety and Pharmacokinetics of SIM0417 Combined With Ritonavir in Healthy Elderly Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM0417-108
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Elder
MeSH Terms: interventions — SIM0417; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIM0417/Ritonavir (Experimental): Single oral dose of 750 mg SIM0417 coadministered with 100 mg ritonavir.
  Interventions: Drug: SIM0417/Ritonavir

INTERVENTIONS:
Drug: SIM0417/Ritonavir — Single oral dose of 750 mg SIM0417 coadministered with 100 mg ritonavir.
  Other Names: 750 mg SIM0417/100 mg ritonavir

SUMMARY:
This is a non-randomized, open-label, single-dose, Phase I clinical study and plans to enroll 12-20 healthy elderly subjects aged 65 and above, including 3-6 subjects aged 75 and above, both men and women.

DETAILED DESCRIPTION:
Each subject will receive SIM0417 combined with ritonavir administration. SIM0417 is single-dose administration, and ritonavir is administered 12 hours before SIM0417 administration (-12hours), at the time of SIM0417 administration (0hour) and 12hours (12hours), SIM0417 is administered under fasting condition, ritonavir is administered under fasting condition either after meal.

The dose of SIM0417 is 750 mg, and the dose of ritonavir is 100 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study content, process, and potential risks of this trial, and voluntarily sign the informed consent.
2. Male and female subjects aged ≥65.
3. Male subjects weigh ≥50 kg, female subjects weigh ≥45 kg; BMI ≥ 19 and ≤ 30 kg/m^2.
4. Subjects of childbearing potential agree to take recognized effective contraceptive measures during the study period and within 1 months after the last dose of the investigational product, starting from signing the informed consent.

Exclusion Criteria:

1. Neurological/psychiatric, respiratory, cardiovascular, gastrointestinal, hematological and lymphatic, endocrine, skeletal-muscular disorders requiring pharmacological intervention or unstable control, hepatic or renal insufficiency, or any other disease or condition that may affect the results of the study or the safety of the subjects.
2. Difficulty in venous blood collection, a history of fainting blood or needles, or those who cannot tolerate blood collection with intravenousindwelling needles.
3. With dysphagia or any history of gastrointestinal diseases that affect drug absorption.
4. Serious infection, trauma, major surgery, gastrointestinal surgery affecting drug absorption within 4 weeks prior to screening
5. Within six months before screening, patients with myocardial infarction, severe/unstable angina pectoris, symptomatic congestive heart failure ( NYHA II-IV ), clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention or clinically significant abnormalities on screening cardiac ultrasound.
6. With blood donation or blood loss was greater than 200 mL within 3 months prior to screening, or blood transfusion or blood products were received within 4 weeks.
7. Have special requirements for diet and cannot comply with the diet provided and corresponding regulations.
8. With specific allergic history ( asthma, urticaria, eczema, etc. ) or allergic constitution ( such as those allergic to two or more drugs, food such as milk, and pollen ) or allergic to any component of the investigational product or investigational product.
9. With special diet ( including pitaya, mango, grapefruit, food or beverage containing caffeine, etc. ) or intense exercise taken within 48 h before the first administration of the investigational product.
10. CYP3A enzyme/P-gp inducer used within 4 weeks prior to screening, or CYP3A enzyme/P-gp inhibitor used within 2 weeks prior to screening; or a prescription drug, over-the-counter drug, herbal medicine was used within 1 week prior to screening; or any health product such as vitamins used during the screening period.
11. Those who have been vaccinated within 1 month before screening (except for the COVID-19 vaccine), or who plan to be vaccinated during treatment / within 2 weeks after the last dose of investigational product.
12. Participation as a subject in any clinical trial with a research intervention within 3 months prior to screening
13. During the first 3 months prior to screening or from the screening period to the first administration period, alcohol was often consumed, i.e., more than 2 units of alcohol per day ( 1 unit = 360 mL beer or 45 mL spirits with 40 % alcohol or 150 mL wine ); or alcohol breath test positive.
14. More than 5 cigarettes per day during the 3 months prior to screening.
15. Have a history of drug abuse or a positive drug abuse screen.
16. At the time of screening or baseline, the blood pressure in the resting state and the pulse are within the following ranges: such as systolic blood pressure <90 mmHg or ≥150 mmHg, diastolic blood pressure <60 mmHg or ≥95 mmHg, pulse <55 bpm or >100 bpm.respiratory rate <12 or >20 breaths/min, SpO2 <95%.
17. Significant abnormalities on ECG at screening (e.g. degree II type II conduction block, left bundle branch block, etc.) QTcF (Fridericia formula) ≥ 470 msec (female)/450 msec (male), or presence of tip-twist Risk factors for ventricular tachycardia (e.g. history of heart failure, family history of prolonged QT interval syndrome)
18. HBV surface antigen, HCV antibody, HIV, or syphilis are positive during screening.
19. Blood biochemical test in following ranges at screening: ALT or AST >1.5 x ULN, triglycerides ≥ 2.3 mmol/L (200 mg/dL), total cholesterol ≥ 6.2 mmol/L (240 mg/dL), blood uric acid ≥ 480 μmol/L (8 mg/dL) Absolute eGFR < 90 mL/min ( eGFR = eGFR（CKD-EPI）× BSA / 1.73).
20. Be positive in SARS-CoV-2 nucleic acid or antigen at screening.
21. Be positive in β-hCG at screening(not applicable to postmenopausal female subjects).

21.Subjects have other conditions that are not suitable for participating in this research, or the subjects may not be able to complete this research for other reasons (judged by the investigator).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Up to 72 hours from SIM0417 administration
  Cmax of SIM0417
AUC0-t | Up to 72 hours from SIM0417 administration
  AUC0-t of SIM0417
AUC0-∞ | Up to 72 hours from SIM0417 administration
  AUC0-∞ of SIM0417
Tmax | Up to 72 hours from SIM0417 administration
  Tmax of SIM0417
t1/2 | Up to 72 hours from SIM0417 administration
  t1/2 of SIM0417
CL/F | Up to 72 hours from SIM0417 administration
  CL/F of SIM0417
Vz/F | Up to 72 hours from SIM0417 administration
  Vz/F of SIM0417

SECONDARY OUTCOMES:
Adverse Events | Up to Day 14
  Proportion of adverse events
Proportion of subjects with abnormal Vital Signs | Up to Day 4
  Proportion of Participants With Clinically Notable Vital Signs
Proportion of subjects with abnormal 12-lead electrocardiogram (ECG) | Up to Day 4
  Proportion of Participants With Clinically Notable ECG
Proportion of subjects with abnormal Laboratory Tests | Up to Day 4
  Proportion of Participants With Clinically Notable Laboratory Tests
Proportion of subjects with abnormal Physical Examination | Up to Day 4
  Proportion of Participants With Clinically Notable Physical Examination

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No